CLINICAL TRIAL: NCT06765720
Title: The Comparison of the Effects of Intermittent Feeding Methods With Nasogastric and Orogastric Tubes on Growth, Nutrition, and Physiological Parameters in Preterm Infants: A Randomized Controlled Trial
Brief Title: Effects of Intermittent Feeding Methods With Nasogastric and Orogastric Tubes in Preterm Infants
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: İstanbul Yeni Yüzyıl Üniversitesi (Other)
Responsible Party: Principal Investigator, Fatma Çarıkçı, Lecturer, İstanbul Yeni Yüzyıl Üniversitesi
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: 20212024BAG-FC
Record Dates: First submitted 2024-12-26; First posted 2025-01-09 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Nasogastric Tube; Orogastric Tube
Keywords: intermittent feeding; enteral feeding; nasogastric tube; orogastric tube; preterm
MeSH Terms: conditions — Premature Birth | interventions — Enteral Nutrition

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intermittent feeding method with nasogastric tube (Experimental): Preterm infants in this group will be fed via a nasogastric tube during the transition period from the initiation of enteral feeding to full oral feeding.
  Interventions: Other: Intermittent feeding method with nasogastric tube
- Intermittent feeding method with orogastric tube (Experimental): Preterm infants in this group will be fed via a orogastric tube during the transition period from the initiation of enteral feeding to full oral feeding.
  Interventions: Other: Intermittent feeding method with orogastric tube

INTERVENTIONS:
Other: Intermittent feeding method with nasogastric tube — 30 Minutes Before Feeding: No invasive procedures will be performed 30 minutes before the daily 1:00 PM feeding.
  5 Minutes Before Feeding: To measure physiological variables, the pulse oximeter probe will be attached to the baby's foot. Oxygen saturation and heart rate will be measured for 2 minutes before feeding.
  Feeding Phase: Measurement values will be taken from the pulse oximeter during feeding.
  Post-Feeding Phase: Any interventions that could affect physiological values will be prevented, and oxygen saturation and heart rate will continue to be measured during the 2-minute period. The baby will be scored using the Early Feeding Skills Assessment Tool.
  Arms: Intermittent feeding method with nasogastric tube
Other: Intermittent feeding method with orogastric tube — 30 Minutes Before Feeding: No invasive procedures will be performed 30 minutes before the daily 1:00 PM feeding.
  5 Minutes Before Feeding: To measure physiological variables, the pulse oximeter probe will be attached to the baby's foot. Oxygen saturation and heart rate will be measured for 2 minutes before feeding.
  Feeding Phase: Measurement values will be taken from the pulse oximeter during feeding.
  Post-Feeding Phase: Any interventions that could affect physiological values will be prevented, and oxygen saturation and heart rate will continue to be measured during the 2-minute period. The baby will be scored using the Early Feeding Skills Assessment Tool.
  Arms: Intermittent feeding method with orogastric tube

SUMMARY:
The study is a randomized controlled, prospective, double-blind trial planned to compare the effects of intermittent feeding methods using nasogastric and orogastric tubes on the growth, nutrition, and physiological parameters of preterm infants.

The population of the study will consist of preterm infants admitted to the Neonatal Intensive Care Unit of a public hospital in Istanbul between February and December 2025. The sample will include 60 preterm infants who meet the research criteria and whose parents agree to participate in the study.

Through randomization, preterm infants will be assigned to either the nasogastric tube group (experimental) or the orogastric tube group (control) from their first enteral feeding until the transition to full oral feeding is completed.

Data for preterm infants in both groups will be collected using the "Preterm Infant Information Form, Early Feeding Skills Assessment Tool, and Nutrition Monitoring Form," which were developed by the researchers based on literature information and expert opinions. These data will encompass growth, nutrition, and physiological parameters before, during, and after feeding throughout the study.

Hypotheses of the Study

H0: There is no significant difference in the effects of intermittent feeding methods using nasogastric and orogastric tubes on growth, feeding complications, and physiological parameters in preterm infants.

H1: There is a significant difference between intermittent feeding methods using nasogastric and orogastric tubes in preterm infants in terms of growth parameters (daily weight gain in grams, time to regain birth weight, time to transition to full enteral feeding, time to transition to full oral feeding, and Early Feeding Skills Assessment Tool score).

H1(1): Preterm infants fed with a nasogastric tube have greater daily weight gain (grams) compared to those fed with an orogastric tube.

H1(2): The time to regain birth weight (days) in preterm infants fed with a nasogastric tube is shorter compared to those fed with an orogastric tube.

H1(3): The time to transition to full enteral feeding (days) in preterm infants fed with a nasogastric tube is shorter compared to those fed with an orogastric tube.

H1(4): The time to transition to full oral feeding (days) in preterm infants fed with a nasogastric tube is shorter compared to those fed with an orogastric tube.

H1(5): The Early Feeding Skills Assessment Tool score of preterm infants fed with a nasogastric tube is higher compared to those fed with an orogastric tube.

H2: There is a significant difference between intermittent feeding methods using nasogastric and orogastric tubes in preterm infants in terms of feeding complications (tube replacement, mucosal trauma, and feeding intolerance).

H2(1): The frequency of tube replacement in preterm infants fed with a nasogastric tube is lower compared to those fed with an orogastric tube.

H2(2): The incidence of mucosal trauma in preterm infants fed with a nasogastric tube is lower compared to those fed with an orogastric tube.

H2(3): The incidence of feeding intolerance in preterm infants fed with a nasogastric tube is lower compared to those fed with an orogastric tube.

H3: There is a significant difference between intermittent feeding methods using nasogastric and orogastric tubes in preterm infants in terms of physiological parameters (oxygen saturation, heart rate, and apnea).

H3(1): The oxygen saturation levels during and after feeding in preterm infants fed with a nasogastric tube are higher compared to those fed with an orogastric tube.

H3(2): The heart rate during and after feeding in preterm infants fed with a nasogastric tube is lower compared to those fed with an orogastric tube.

H3(3): The incidence of apnea in preterm infants fed with a nasogastric tube is lower compared to those fed with an orogastric tube.

DETAILED DESCRIPTION:
Enteral feeding is preferred as a safe method for preterm infants whose oral feeding skills have not yet developed or who are not ready for oral feeding. It is also implemented to support intestinal development and avoid the long-term side effects of parenteral nutrition. Enteral feeding is a method that allows infants to receive nutrients by utilizing the natural functions of their gastrointestinal system through the advancement of a feeding tube from the mouth or nose to the stomach. Feeding via nasogastric and orogastric tube methods, commonly used in neonatal intensive care units, provides enteral nutrition support for preterm infants. The nasogastric tube is inserted through the nose into the stomach, while the orogastric tube is placed through the mouth into the stomach. Both feeding methods offer various advantages and disadvantages based on the individual needs and clinical conditions of the infants. Therefore, the selection of the feeding method should involve a comprehensive evaluation of the potential benefits and risks unique to each method for the infant.

Since preterm infants breathe nasally, feeding with a nasogastric tube can cause partial nasal obstruction, leading to increased airway resistance and respiratory workload. This situation may result in the collapse of the pharyngeal airways and an increased incidence of apnea of prematurity in preterm infants. Additionally, prolonged feeding with a nasogastric tube in preterm infants has been reported to cause nasal septum defects. In contrast, while the placement and fixation of orogastric tubes are generally easier, these tubes can lead to complications such as displacement or incorrect placement into the lungs, aspiration, increased respiratory resistance, and bradycardia episodes due to vagal stimulation. Furthermore, the prolonged use of orogastric tubes in very low birth weight preterm infants may increase the risk of palate deformation. Therefore, the selection of the feeding method should be based on the infant's health status, respiratory functions, and other clinical parameters.

In the literature, studies investigating the effects of nasogastric and orogastric tubes on preterm infants have shown that the sample groups are limited, crossover designs were used, and there are methodological limitations regarding the determination of evaluation parameters and the process of transition to full enteral feeding. It has been observed that there is a need for a randomized controlled study with a large sample size to examine the effects of intermittent feeding methods using nasogastric and orogastric tubes on the growth, nutrition, and physiological parameters of preterm infants. Accordingly, this research was planned as a randomized controlled, prospective, double-blind study to compare the effects of intermittent feeding methods using nasogastric and orogastric tubes on the growth, nutrition, and physiological parameters of preterm infants.

The infants to be included in the study will be selected according to the determined inclusion criteria and then randomly divided into two groups: nasogastric tube feeding group and orogastric tube feeding group.

In the study, the randomization process will be carried out using the urn method. The urn method is equivalent to complete randomization and will be expressed with two parameters, α and β. These parameters will be symbolized as balls in red and white colors. White or red color will represent α; β will represent the opposite color of α. In each assignment process, the color of a randomly selected ball will determine which group the infant will be assigned to: when a white ball is selected, the infant will be assigned to the orogastric group, and when a red ball is selected, the infant will be assigned to the nazogastric group. In the study, the white ball will be designated as the orogastric group, and the red ball will be designated as the nazogastric group. For each new infant participant who meets the sample criteria, the previously prepared balls will be stored in a black bag, and a nurse on duty in the unit will randomly select one with their eyes closed. Based on the color of the selected ball, infants will be assigned to the groups, ensuring a random distribution between groups

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants with a gestational age of ≥30 weeks at birth, determined according to the mother's last menstrual period, and appropriate for gestational age,
* Postmenstrual age of ≥30 weeks at the time of inclusion in the study,
* Recommended for enteral feeding by a neonatologist,
* Infants starting enteral feeding for the first time and fed at three-hour intervals using gravity-assisted nasogastric or orogastric tubes,
* Infants who have not undergone oral feeding trials,
* Infants who have not received any oral motor interventions,
* Infants whose parents have given consent for inclusion in the study and signed an informed consent form after being provided with detailed information.

Exclusion Criteria:

* Infants receiving mechanical ventilation support during the study,
* Infants with an umbilical catheter,
* Infants who received intubation, CPAP, or nasal prong oxygen support for more than 14 days before inclusion in the study,
* Infants with craniofacial anomalies such as cleft palate, cleft lip, or facial muscle paralysis,
* Infants with any gastrointestinal, neurological, or chromosomal disease (e.g., necrotizing enterocolitis, grade III and IV intracranial hemorrhage, periventricular leukomalacia, hydrocephalus, Down syndrome, and other diseases),
* Infants with severe bronchopulmonary dysplasia according to the criteria of Jobe and Bancalari (2001) or requiring surgical treatment for patent ductus arteriosus.

Ages: 30 Weeks to 36 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Time to transition to full enteral feeding | From the infant's birth until the time they achieve full enteral feeding.Time frame is through study completion, an average of 8 months.
  An infant will be considered to have transitioned to full enteral feeding once all energy and nutrient needs are met for 48 hours through intermittent enteral feeding eight times a day at three-hour intervals.
Time to transition to full oral feeding | From the infant's birth until the time they achieve full oral feeding.Time frame is through study completion, an average of 8 months.
  An infant will be considered to have achieved full oral feeding once they can take 8 feedings per day orally at three-hour intervals for 48 hours and gain 20-30 g/kg.
Time to regain birth weight | The number of days it takes for them to recover the weight they lost after birth.Time frame is through study completion, an average of 8 months.
Daily weight gain | It will be measured every day throughout the research. Time frame is through study completion, an average of 8 months.
Early Feeding Skills Assessment Tool score | It will be evaluated every day throughout the research.Time frame is through study completion, an average of 8 months.

SECONDARY OUTCOMES:
Frequency of tube changes | It will be evaluated every day throughout the research.Time frame is through study completion, an average of 8 months.
Incidence of mucosal trauma | It will be evaluated every day throughout the research.Time frame is through study completion, an average of 8 months.
Development and frequency of feeding intolerance | Time frame is through study completion, an average of 8 months.
Oxygen saturation levels | Time frame is through study completion, an average of 8 months.
Heart rate variability | Time frame is through study completion, an average of 8 months.
Incidence of apnea | Time frame is through study completion, an average of 8 months.

CONTACTS AND LOCATIONS:
Overall Officials: Burcu Aykanat Girgin, Assoc. Dr., Study Director — Saglik Bilimleri Universitesi
Locations (1):
- Yeni Yüzyıl University, Zeytinburnu, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No